CLINICAL TRIAL: NCT02397707
Title: A Phase 1 Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Pharmacokinetics of GS-9857 in Subjects With Normal Hepatic Function and Moderate or Severe Hepatic Impairment
Brief Title: Pharmacokinetics of Voxilaprevir in Adults With Normal Hepatic Function and Moderate or Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-338-1126; 2015-000342-30 (EudraCT Number)
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — voxilaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Hepatic Impaired (Experimental): Participants with moderate hepatic impairment and matched healthy controls will receive a single dose of voxilaprevir on Day 1.
  Interventions: Drug: Voxilaprevir
- Severe Hepatic Impaired (Experimental): Participants with severe hepatic impairment and matched healthy controls will receive a single dose of voxilaprevir on Day 1.
  Interventions: Drug: Voxilaprevir

INTERVENTIONS:
Drug: Voxilaprevir — 100 mg tablet administered orally
  Other Names: GS-9857

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of a single dose of voxilaprevir (formerly GS-9857) in participants with normal hepatic function, moderate hepatic impairment and severe hepatic impairment. Participants in the healthy control group will be matched to participants with impaired hepatic function by gender, age (± 10 years), and body mass index (± 15%).

ELIGIBILITY:
Key Inclusion Criteria:

* All individuals:

  * Screening laboratory values within defined thresholds for group
  * Use of two effective contraception methods if female of childbearing potential or sexually active male
* For individuals with moderate hepatic impairment:

  * Diagnosis of chronic (> 6 months) hepatic impairment
  * Score on the Child-Pugh-Turcotte (CPT) scale of 7-9 at screening (Child Pugh Class B).
* For individuals with severe hepatic impairment:

  * Diagnosis of chronic (> 6 months) hepatic impairment
  * Score on the CPT scale of 10-15 at screening (Child Pugh Class C)
* For individuals with normal hepatic function:

  * Hepatitis C Virus (HCV) antibody and hepatitis B surface antigen negative

Key Exclusion Criteria:

* All individuals:

  * Pregnant or nursing female or male with pregnant female partner
  * HIV infection
  * History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment or compliance with the protocol
* For individuals with moderate or severe hepatic impairment:

  * Active HCV infection
  * Current hepatic encephalopathy
  * Variceal bleeding in the last 6 months unless banded
  * Prior placement of a portosystemic shunt
  * History of hepatorenal or hepatopulmonary syndrome
  * Spontaneous bacterial peritonitis currently or within the last 6 months
  * Hospitalization within the last 2 months related to cirrhosis
  * Confirmed hypotension
  * Suspicion of hepatocellular carcinoma

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2016-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas
- APEX GmbH, München, Germany
- Auckland Clinical Studies, Auckland, New Zealand

REFERENCES:
- [Result] Lawitz E, Marbury T, Kirby BJ, Au NT, Mathias A, Stamm LM, et al. The Effect of Renal or Hepatic Impairment on the Pharmacokinetics of GS-9857, A Pan-Genotypic HCV NS3/4A Protease Inhibitor [Abstract FRI-167]. J Hepatology 2016:S613-S4.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, Germany, and New Zealand. The first participant was screened on 24 March 2015. The last study visit occurred on 04 March 2016.
Pre-assignment Details: 54 participants were screened. 33 participants were enrolled, 14 participants with normal hepatic function, 10 with Moderate Hepatic Impairment (MHI), and 9 with Severe Hepatic Impairment (SHI). Five of the same participants with normal hepatic function served as matched controls for the MHI and SHI Arms/Groups.
Groups:
- Normal Hepatic Function: Participants with normal hepatic function received single dose of voxilaprevir 100 mg tablet orally on Day 1.
- Moderate Hepatic Impairment (MHI): Participants with moderate hepatic impairment received single dose of voxilaprevir 100 mg tablet orally on Day 1.
- Severe Hepatic Impairment (SHI): Participants with severe hepatic impairment received single dose of voxilaprevir 100 mg tablet orally on Day 1.
Period: Overall Study
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment (MHI) | Severe Hepatic Impairment (SHI)
Started | 14 | 10 | 9
Completed | 14 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment (MHI) | Severe Hepatic Impairment (SHI) | Total
Number analyzed (Participants) | 14 | 10 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9.8) | 55 (6.7) | 55 (7.0) | 54 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 11
  Male | 9 | 6 | 7 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Black | 3 | 1 | 0 | 4
  Native Hawaiian or Pacific Islander | 1 | 1 | 0 | 2
  White | 9 | 8 | 9 | 26
  Not Permitted | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 5 | 15
  Not Hispanic or Latino | 7 | 7 | 4 | 18
  Not Permitted | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 6 | 25
  New Zealand | 3 | 2 | 1 | 6
  Germany | 0 | 0 | 2 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (2.21) | 27.6 (3.90) | 28.4 (3.86) | 27.8 (3.18)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter of Voxilaprevir: AUClast
Description: AUClast is defined as the area under the plasma concentration versus time curve from time zero to the last quantifiable concentration. Data presented are unadjusted geometric means and confidence intervals.
Time Frame: 0 (pre-dose ≤ 5 minutes), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours post-dose
Population: PK Analysis Set included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value reported by the PK laboratory for the corresponding analyte. Five of the same participants with normal hepatic function served as matched controls for the MHI and SHI Arms/Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Groups:
- Normal Hepatic Function (Matched Control for MHI): Normal Hepatic Function (matched control for MHI) included participants that served as controls for participants with MHI.
- Normal Hepatic Function (Matched Controls for SHI): Normal hepatic function (matched controls for SHI) included participants that served as controls for participants with SHI.
Arm/Group | Moderate Hepatic Impairment (MHI) | Severe Hepatic Impairment (SHI) | Normal Hepatic Function (Matched Control for MHI) | Normal Hepatic Function (Matched Controls for SHI)
Number analyzed (Participants) | 10 | 9 | 10 | 9
h*ng/mL | 2058.5 [1034 to 4098.1] | 3872.5 [2173.1 to 6901.2] | 500.1 [307 to 814.6] | 601.2 [372.8 to 969.6]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (MHI) vs Normal Hepatic Function (Matched Control for MHI); An analysis of variance (ANOVA) appropriate for a parallel design was fitted to the natural logarithmic transformation of voxilaprevir AUClast. A 90% confidence interval (CI) was constructed for the geometric least squares mean (GLSM) ratio of AUClast for the comparison groups using two 1-sided tests; Test type: Other; Geometric Least-Square Mean (GLSM)Ratio% = 411.62, 90% CI 2-sided [214.72 to 789.08]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment (SHI) vs Normal Hepatic Function (Matched Controls for SHI); An ANOVA appropriate for a parallel design was fitted to the natural logarithmic transformation of voxilaprevir AUClast. A 90% CI was constructed for the GLSM ratio of AUClast for the comparison groups using two 1-sided tests; Test type: Other; GLSM Ratio (%) = 644.15, 90% CI 2-sided [364.67 to 1137.82]

2. Primary Outcome: PK Parameter of Voxilaprevir: AUCinf
Description: AUCinf is defined as the area under the plasma concentration versus time curve extrapolated to infinite time. Data presented are unadjusted geometric means and confidence intervals.
Time Frame: 0 (pre-dose ≤ 5 minutes), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours postdose
Population: Participants in the PK Analysis Set were analyzed. Five of the same participants with normal hepatic function served as matched controls for the MHI and SHI Arms/Groups.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Moderate Hepatic Impairment (MHI) | Severe Hepatic Impairment (SHI) | Normal Hepatic Function (Matched Control for MHI) | Normal Hepatic Function (Matched Controls for SHI)
Number analyzed (Participants) | 10 | 9 | 10 | 9
h*ng/mL | 2227.1 [1122 to 4420.7] | 4107.5 [2331.7 to 7235.7] | 557.8 [351.8 to 884.6] | 685 [426.1 to 1101.2]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (MHI) vs Normal Hepatic Function (Matched Control for MHI); An ANOVA appropriate for parallel design was fitted to the natural logarithmic transformation of voxilaprevir AUCinf. A 90% CI was constructed for the GLSM ratio of AUClast for the comparison groups using two 1-sided tests; Test type: Other; GLSM Ratio (%) = 399.24, 90% CI 2-sided [210.89 to 755.81]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment (SHI) vs Normal Hepatic Function (Matched Controls for SHI); An ANOVA appropriate for parallel design was fitted to the natural logarithmic transformation of voxilaprevir AUCinf. A 90% CI was constructed for the GLSM ratio of AUCinf for the comparison groups using two 1-sided tests; Test type: Other; GLSM Ratio (%) = 599.63, 90% CI 2-sided [342.36 to 1050.22]

3. Primary Outcome: PK Parameter of Voxilaprevir: Cmax
Description: Cmax is defined as the maximum observed plasma concentration of drug.Data presented are unadjusted geometric means and confidence intervals.
Time Frame: 0 (pre-dose ≤ 5 minutes), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment (MHI) | Severe Hepatic Impairment (SHI) | Normal Hepatic Function (Matched Control for MHI) | Normal Hepatic Function (Matched Controls for SHI)
Number analyzed (Participants) | 10 | 9 | 10 | 9
ng/mL | 189.7 [85.2 to 422.3] | 370.8 [183.6 to 749] | 56.1 [38.2 to 82.2] | 51.9 [35.1 to 76.9]
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment (MHI) vs Normal Hepatic Function (Matched Control for MHI); An ANOVA appropriate was fitted to the natural logarithmic transformation of voxilaprevir Cmax. A 90% CI was constructed for the GLSM ratio of AUClast for the comparison groups using two 1-sided tests; Test type: Other; GLSM Ratio (%) = 338.41, 90% CI 2-sided [168.96 to 677.79]
Statistical Analysis 2: Comparison: Severe Hepatic Impairment (SHI) vs Normal Hepatic Function (Matched Controls for SHI); [analysis description as in outcome 3, analysis 1]; Test type: Other; GLSM Ratio (%) = 713.92, 90% CI 2-sided [384.07 to 1327.06]

ADVERSE EVENTS:
Time Frame: First dose date up to 31 days
Description: Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment (MHI) | Severe Hepatic Impairment (SHI)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 2/14 | 3/10 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (N=14) | Moderate Hepatic Impairment (MHI) (N=10) | Severe Hepatic Impairment (SHI) (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years